CLINICAL TRIAL: NCT00607841
Title: A Phase I/II Non-Randomized, Open-Label, Dose-Finding Study of Ispinesib (SB-715992) Followed By a Fixed-Dose Study in Chemotherapy-Naïve Patients With Metastatic Breast Cancer (MBC).
Brief Title: A Study of Ispinesib in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial stopped for administrative reasons prior to official determination of MTD.
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CY 3121
Record Dates: First submitted 2008-01-22; First posted 2008-02-06 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — ispinesib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Escalation Cohort 1 (Experimental): Ispinesib given on days 1 and 15 of a 28 day cycle.
  Interventions: Drug: Ispinesib
- Dose Escalation Cohort 2 (Experimental): Ispinesib given on days 1 and 15 of a 28 day cycle.
  Interventions: Drug: Ispinesib
- Dose Escalation Cohort 3 (Experimental): Ispinesib given on days 1 and 15 of a 28 day cycle.
  Interventions: Drug: Ispinesib

INTERVENTIONS:
Drug: Ispinesib — 10 mg/m2 dose as a 1-hour intravenous infusion.
  Other Names: SB-715992
  Arms: Dose Escalation Cohort 1
Drug: Ispinesib — 12 mg/m2 dose as a 1-hour intravenous infusion.
  Other Names: SB-715992
  Arms: Dose Escalation Cohort 2
Drug: Ispinesib — 14 mg/m2 dose as a 1-hour intravenous infusion.
  Other Names: SB-715992
  Arms: Dose Escalation Cohort 3

SUMMARY:
The Phase I portion was a dose-escalation study designed to assess safety and tolerability in patients with metastatic breast cancer. Phase II was intended to measure response rate in patients with metastatic breast cancer but did not enroll because the Phase I portion was halted prior to Maximum Tolerated Dose (MTD) determination.

DETAILED DESCRIPTION:
Only the Phase I portion of the study was enrolled. The Phase I dose-escalation portion of the trial was designed to determine the Dose Limiting Toxicities (DLT) and MTD of Ispinesib (SB-715992) monotherapy when administered as a one-hour infusion on Days 1 and 15 of a 28-day cycle in female patients with locally advanced or metastatic breast cancer. The Phase II regimen was intended to evaluate the MTD determined in Phase I in chemotherapy-naïve female patients with measurable, locally advanced or metastatic breast cancer. Phase II was intended to assess the overall response rate (ORR) derived from individual patient assessments of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) based on RECIST, as determined by independent review.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced (Stage IIIb) or metastatic (Stage IV) adenocarcinoma of the breast. Staging is determined according to the American Joint Committee on Cancer, Cancer Staging Manual, Sixth Edition
2. Has not received prior cytotoxic chemotherapy for breast cancer and is not currently receiving other anti-cancer therapy, including trastuzumab or other cytostatics, hormonal therapy, radiotherapy, immunotherapy, biologic or investigational agent(s).

   Note: Prior therapy does not include (a) previous surgery and/or radiotherapy (if less than 25% of pelvic bone marrow), (b) adjuvant and/or palliative hormonal therapy, (c) gefitinib (Iressa®) or trastuzumab (Herceptin®) given as monotherapy.
3. Phase I only: Patients who have previously received anthracycline therapy in either the adjuvant or neoadjuvant setting may participate, provided a minimum of one year has elapsed since last treatment.
4. Phase I only: Must have evaluable, but not necessarily measurable disease by imaging.
5. Phase II only: Must have at least one unidimensionally measurable lesion evaluable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. The lesion(s) must be documented by photography, radiography, direct measurement, or palpation.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
7. Female patients, 18 years of age or older.
8. A female is eligible to enter and participate in the study if she is of:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:

      * Has had a hysterectomy,
      * Has had a bilateral oophorectomy (ovariectomy),
      * Has had a bilateral tubal ligation, or
      * Is post-menopausal (a demonstration of total cessation of menses for ≥ 1 year.
   2. Childbearing potential, has a negative serum pregnancy test at screening, and agrees to one of the following:

      * Intrauterine Device (IUD),
      * Vasectomized partner who is sterile prior to the female patient's entry and is the sole sexual partner for that female,
      * Complete abstinence from sexual intercourse for two weeks before exposure to investigational product, throughout the clinical trial, and for at least one week after the last dose of investigational product, or
      * Double barrier contraception (condom with spermicidal jelly, foam, suppository, or film, diaphragm with spermicide, or male condom and diaphragm).
      * Progesterone based contraceptive with a failure rate of < 1%.
9. A signed and dated written informed consent is obtained from the patient or the patient's legally acceptable representative prior to screening.

Exclusion Criteria:

1. Receipt of prior cytotoxic chemotherapy except in an adjuvant or neo adjuvant setting
2. Has not recovered from prior therapy including any major surgery, radiotherapy, immunotherapy, biologic or investigational agent(s).
3. Absolute neutrophil count (ANC) <1,500/mm3.
4. Platelets < 100,000/mm3.
5. Creatinine clearance ≤ 40 mL/min as calculated by the Cockcroft-Gault Formula.
6. Total bilirubin greater than or equal to 1.5 x ULN
7. Alanine aminotransferase (ALT) greater than 2 times the upper limit of normal (ULN) in the absence of liver metastases (patients with serum transaminase levels up to 5 times ULN in the presence of liver metastases may be enrolled following approval by Cytokinetics Medical Monitor).
8. Alkaline Phosphate (ALP) greater than or equal to 5 x ULN
9. Female patients who are pregnant or lactating.
10. Women of reproductive potential who do not agree to use an effective contraceptive method.
11. Any unstable, pre-existing major medical condition or history of other malignancies (except excised cervical or basal skin/squamous cell carcinoma).
12. Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol.
13. Evidence of central nervous system (CNS) metastases or leptomeningeal disease
14. Evidence of any other malignancy
15. Previous exposure to any Investigational Agent
16. Radiation therapy within 28 days, or within 3 months if blood urea nitrogen (BUN) is ≥20mg/dl

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity and Maximum Tolerated Dose of ispinesib administered as a 1-hr intravenous infusion on Day 1 of a 28-day cycle in female patients with Stage IIIB or IV breast cancer | 28 days
Dose Limiting Toxicity and Maximum Tolerated Dose of ispinesib administered as a 1-hr intravenous infusion on Day 15 of a 28-day cycle in female patients with Stage IIIB or IV breast cancer | 28 days
Assessment of response rate based on Response Evaluation Criteria in Solid Tumors (RECIST) in patients with metastatic breast cancer | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Wolff, MD, FACC, Study Chair — Cytokinetics
Locations (3):
- Peru (3):
  - Hospital Nacional Alberto Sabogal Sologúren, Lima
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Instituto Nacional de Enfermedades Neoplásicas, Lima